CLINICAL TRIAL: NCT03286569
Title: Study the Effect of Upper Expansion Appliances on Lower Jaw Forward Projection/Growth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00001731
Record Dates: First submitted 2015-04-12; First posted 2017-09-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Overbite (Excessive) Horizontal
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active upper Wilson appliance (Active Comparator): Active upper arch Wilson quadhelex appliance
  Interventions: Device: Upper arch Wilson quadhelex appliance
- Non active upper expansion appliance (Placebo Comparator): Non-Active upper arch Wilson quadhelex appliance
  Interventions: Device: Upper arch Wilson quadhelex appliance

INTERVENTIONS:
Device: Upper arch Wilson quadhelex appliance — Upper arch Wilson quadhelex appliance

SUMMARY:
Young children with backward positioned lower jaw/chin will be recruited to have an upper jaw expansion appliance. Previous research showed that the use of similar appliances can lead to lower jaw forward growth. 60 young children aged 9-11 will be recruited to have either active or non-active Wilson type upper arch expansion appliance. Patients will have special x-ray (Cone Beam computed tomography) before and after treatment (after 9 months) of starting the treatment. After participation, routine orthodontic treatment will be continued.

DETAILED DESCRIPTION:
Previous research showed that the use of upper jaw expansion appliances can lead to lower jaw forward growth (1). 60 young children aged 9-11 with backward positioned lower jaw/chin will be recruited to have either active or non-active Wilson type upper arch expansion appliance. Patients will have special x-ray (Cone Beam computed tomography) before and after treatment (after 9 months) of starting the treatment. After participation, routine orthodontic treatment will be continued.

ELIGIBILITY:
Inclusion Criteria:

1. Class II skeletal due to lower jaw backward projection
2. Class II malocclusion
3. Early mixed dentition (all first permanent molars erupted, as well as all erupting upper and lower permanent incisors)

Exclusion Criteria:

1. Other orthodontic treatment provided
2. Growth problems (craniofacial syndromes, etc.)

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Lower jaw size | 9 months
  Lower jaw size will be evaluated by computed tomography.
Lower jaw projection | 9 months
  Lower jaw projection will be evaluated by computed tomography.

SECONDARY OUTCOMES:
Jaw joint size | 9 months
  Jaw joint size will be evaluated by CBCT
Base of skull bone size | 9 months
  Base of skull bone size will be evaluated by CBCT
Base of skull bone position | 9 months
  Base of skull bone positions will be evaluated by CBCT
Jaw joint position | 9 months
  Jaw joint will be evaluated by CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Result] McNamara JA Jr, Sigler LM, Franchi L, Guest SS, Baccetti T. Changes in occlusal relationships in mixed dentition patients treated with rapid maxillary expansion. A prospective clinical study. Angle Orthod. 2010 Mar;80(2):230-8. doi: 10.2319/040309-192.1. PMID 19905846
- [Result] Guest SS, McNamara JA Jr, Baccetti T, Franchi L. Improving Class II malocclusion as a side-effect of rapid maxillary expansion: a prospective clinical study. Am J Orthod Dentofacial Orthop. 2010 Nov;138(5):582-91. doi: 10.1016/j.ajodo.2008.12.026. PMID 21055598